CLINICAL TRIAL: NCT00438191
Title: A Clinical Trial of Full Time vs. As Needed Splint Wear for DeQuervain's Tenosynovitis
Brief Title: A Clinical Trial of Splinting for DeQuervain's Tenosynovitis
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Principal Investigator; Director of Research, Hand Service, Massachusetts General Hospital
Other Study IDs: 2005-P-002319
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: DeQuervain's Tenosynovitis
Keywords: DeQuervain's tenosynovitis; splinting; grip strength; satisfaction; DASH questionnaire
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: Subjects who wear the splint whenever the feel the need.
- 2: Subjects who wear the splint whenever possible.

SUMMARY:
DeQuervain's tenosynovitis is characterized by pain on the pain on the radial (thumb) side of the wrist problems with thumb function. At this point, the standard care is to change daily activities, use a thumb brace, and the possible use of painkillers. There is a difference in opinion among physical therapists about how to use the splint in the treatment of DeQuervain tenosynovitis. Some physicians tell patients to wear the brace at all times while other therapists encourage patients to exercise and use the brace as needed. Both approaches to using the splint are accepted as standard. The purpose of this study is to test and evaluate these two ways of splinting and assess which one is better for patients with DeQuervain tenosynovitis.

DETAILED DESCRIPTION:
De Quervain's tenosynovitis (stenosing tenosynovitis of the first dorsal extensor compartment) is characterized by pain on the radial (thumb) side of the wrist and impairment of thumb and wrist function. Histological evaluation is consistent with a chronic rather than an acute tenosynovitis consistent with the often prolonged course of this disease.

Nonoperative treatments include modification of activities, splint immobilization, icing and anti-inflammatory medication, and corticosteroid injections. Long opponens splinting (or short arm thumb spica splinting; a splint that immobilizes the wrist and the thumb) is standard and well accepted. There is no consensus on the best protocol for use of the splint. Some authors advocate full time splinting for 4 - 6 weeks, with the rationale that tendonitis will resolve with strict rest. Other authors, perhaps aware of histological evidence that De quervain's is a chronic rather than acute inflammatory condition, feel that the splint serves merely to relieve symptoms and is best used as best suits each individual patient. To our knowledge, there are not data available regarding these disparate views.

The ultimate prognosis for recovery in the condition seems satisfying, regardless of the treatment, and spontaneous recovery is the rule. Psychological and personality factors, such as pain anxiety, catastrophizing, and depression are strongly related to upper extremity specific health status and may also influence recovery.

The primary goal of this study is to determine which protocol of splinting leads to better outcome in non-surgical treatment of DeQuervain's tenosynovitis. As a secondary goal and to generate hypotheses for later studies we would like to evaluate the influence of psychosocial factors on both objective (grip strength) and subjective (DASH questionnaire) measures of outcome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age 18 years or greater)
* Physician very confident about the diagnosis of DeQuervain's tenosynovitis.

Exclusion Criteria:

* Patients with previous history of surgical treatment for De Quervain's.
* Skin conditions making splint wear problematic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the MGH Hand and Upper Extremity Service.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2005-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- As-Desired Splinting: Subjects who wear the splint as desired
- Full Time Splinting: Subjects who wear the splint as much as possible
Period: Overall Study
Arm/Group | As-Desired Splinting | Full Time Splinting
Started | 43 | 40
Completed | 32 | 26
Not Completed | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | As-Desired Splinting | Full Time Splinting | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.93 (14.58) | 48.74 (13.90) | 49.26 (14.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  United States | 43 | 40 | 83
Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire [Mean (Standard Deviation); unit: units on a scale] — The DASH questionnaire measures the upper extremity disability on a scale from 0-100, 0 is no disability and 100 is the most disability.
  units on a scale | 36.5 (19.0) | 33.3 (17.8) | 34.96 (18.40)
Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Pain intensity was measured using the Numeric Rating Scale, on a scale from 0-10, where 0 is no pain and 10 is the most pain.
  units on a scale | 5.5 (2.3) | 5.8 (2.4) | 5.6 (2.4)
Center for Epidemiologic Studies Depression Scale - Revised (CES-D) [Mean (Standard Deviation); unit: units on a scale] — The CESD-R measures symptom of depression in nine different groups. The range of possible scores is between 0 (for those who say 'not at all or less than one day to all 20 questions) and 60 (nearly everyday for 2 weeks for all 20 questions).
  units on a scale | 16.3 (6.5) | 16.3 (8.7) | 16.3 (7.6)
Pain Catastrophizing scale (PCS) [Mean (Standard Deviation); unit: units on a scale] — The Pain Catastrophizing Scale measures a set of mal-adaptive cognitive conditions while in pain. The score ranges from 0-52, ranging from least to most catastrophic thinking.
  units on a scale | 20.9 (8.7) | 17.5 (9.5) | 19.3 (9.2)
Grip Strength [Mean (Standard Deviation); unit: percentage of non-affected hand] — Grip strength measured as a percentage of the non-affected hand.
  percentage of non-affected hand | 54.1 (22.9) | 58.6 (18.7) | 56.3 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire
Description: The DASH questionnaire measures upper extremity disability on a scale from 0-100, where 0 is no disability and 100 is severe disability.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | As-Desired Splinting | Full Time Splinting
Number analyzed (Participants) | 32 | 26
units on a scale | 28 (15) | 29 (20)

2. Secondary Outcome: Grip Strength
Description: Grip strength is measured as a percentage of the non-affected or least affected side.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of non-affected hand
Arm/Group | As-Desired Splinting | Full Time Splinting
Number analyzed (Participants) | 32 | 26
percentage of non-affected hand | 86 (25) | 87 (18)

3. Secondary Outcome: Treatment Satisfaction
Description: Treatment satisfaction was measured on a scale from 0-10, where 0 is complete dissatisfaction and 10 is complete satisfaction
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | As-Desired Splinting | Full Time Splinting
Number analyzed (Participants) | 32 | 26
units on a scale | 6.3 (2.6) | 6.4 (2.9)

4. Secondary Outcome: Pain Intensity
Description: Pain intensity was measured using the Numeric Rating Scale, on a scale from 0-10, where 0 is no pain and 10 is the most pain.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | As-Desired Splinting | Full Time Splinting
Number analyzed (Participants) | 32 | 26
units on a scale | 3.8 (2.0) | 4.4 (2.9)

ADVERSE EVENTS:
Arm/Group | As-Desired Splinting | Full Time Splinting
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/40
Other Adverse Events (participants affected / at risk) | 0/43 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes